CLINICAL TRIAL: NCT04901650
Title: Pain Prevalence in Hospitalized Patients in Hospital Universitario de Gran Canaria Doctor Negrín
Brief Title: Pain Prevalence in Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, Ángel Becerra, Principal Investigator, Dr. Negrin University Hospital
Other Study IDs: PainPrevalence
Record Dates: First submitted 2021-05-17; First posted 2021-05-25 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Pain
Keywords: Pain prevalence; Pain management; Opioids; Non-steroidal antiinflamatory drugs
MeSH Terms: conditions — Pain; Agnosia | interventions — Fertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inpatient population: A survey will be administered to find out the prevalence of pain in hospitalized patients for any cause and its intensity. The medical history will be reviewed to assess the presence of pain medications and their impact on the pain perception and patients' satisfaction.
  Interventions: Diagnostic Test: Survey

INTERVENTIONS:
Diagnostic Test: Survey — A survey will be administered to find out the prevalence of pain in hospitalized patients for any cause and its intensity. The medical history will be reviewed to assess the presence of pain medications and their impact on the pain perception and patients' satisfaction.

SUMMARY:
Pain is a sensation of discomfort, annoyance or distress, described as an unpleasant subjective sensory and emotional experience associated with actual or potential injury, and may associate vegetative, psychological, emotional, and behavioral responses. It is the main reason for medical consultation and in many cases it is assumed as inevitable. It is also a clinical symptom and generates negative consequences. As a result, people who suffer from "pain" may see their quality of life diminished.

On many occasions, either due to the high healthcare burden, because pain is not the reason for consultation or because the main pathology suffered by the patient is not the cause of the pain, not attention is given to it.

The objective of this study is to evaluate the prevalence of pain in the inpatient population, analyzing its presence and intensity in patients admitted to the Doctor Negrín University Hospital of Gran Canaria. Likewise, it is interesting to know what percentage of patients with pain have analgesics and the degree of relief with the treatment received. As a secondary objective, it is intended to establish whether there is a relationship between factors dependent on the patient and the presence of pain.

DETAILED DESCRIPTION:
Pain is a sensation of discomfort, annoyance or distress, described as an unpleasant subjective sensory and emotional experience associated with actual or potential injury, and may associate vegetative, psychological, emotional, and behavioral responses. It is the main reason for medical consultation and in many cases it is assumed as inevitable. It is also a clinical symptom and generates negative consequences. As a result, people who suffer from "pain" may see their quality of life diminished.

Its appearance requires a multidisciplinary treatment, from different perspectives and through different mechanisms, taking into account the individual characteristics of each patient; since this symptom can be modified which today are not strictly described.

On many occasions, either due to the high healthcare burden, because pain is not the reason for consultation or because the main pathology suffered by the patient is not the cause of the pain, not attention is given to it.

It is necessary to carry out a good questionnaire to the patient and take into account the presence or absence of pain, regardless of the primary pathology that concerns us, in order to be able to provide correct attention. Pain control may greatly vary the patient's vision of his ailment and with it, his psycho-emotional state, his attitude and his collaboration, reducing the impact on his quality of life and the duration of hospital admission.

The objective of this study is to evaluate the prevalence of pain in the inpatient population, analyzing its presence and intensity in patients admitted to the Doctor Negrín University Hospital of Gran Canaria. Likewise, it is interesting to know what percentage of patients with pain have analgesics and the degree of relief with the treatment received. As a secondary objective, it is intended to establish whether there is a relationship between factors dependent on the patient and the presence of pain.

ELIGIBILITY:
Inclusion Criteria:

* hospital admission for more than 24 hours
* age >18 years old
* desire and express authorization of the individual to participate in the study by accepting informed consent

Exclusion Criteria:

* refusal of the subject to participate in the study
* alterations in cognitive status, speech or comprehension problems
* language barrier
* psychiatric pathology
* Covid patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for more than 24 hours will be surveyed at the same date.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Pain Prevalence | 24 hours throughout the hospital admission
  Pain prevalence will be obtained from patients who have been hospitalized for more than 24 hours at the Hospital.

SECONDARY OUTCOMES:
Patient satisfaction assessed by VAS (from 0 to 10) | 24 hours throughout the hospital admission
  Satisfaction regarding the pain management will be obtained from patients who have been hospitalized for more than 24 hours at the Hospital using a Visual Analogue Scale from 0 to 10.
Percentage of patients receiving drugs for pain management | 24 hours throughout the hospital admission
  Pain management will be evaluated reviewing the medical history from patients who have been hospitalized for more than 24 hours at the Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Aurelio Rodríguez-Pérez, PhD, Study Chair — Hospital Universitario de Gran Canaria Doctor Negrín
Locations (1):
- Ángel Becerra, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared as request to the Principal Investigator